CLINICAL TRIAL: NCT02275286
Title: Phase I-II Prospective Trial, Multicenter, Open Label, Exploring the Combination of Trabectedin Plus Radiotherapy in Soft Tissue Sarcoma Patients
Brief Title: Trabectedin Plus Radiotherapy in Soft Tissue Sarcoma Patients
Acronym: TRASTS
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Grupo Espanol de Investigacion en Sarcomas (Other)
Collaborators: Centre Leon Berard (Other); Italian Sarcoma Group (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEIS 37
Record Dates: First submitted 2014-10-17; First posted 2014-10-27 (Estimated); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Liposarcoma, Myxoid; Sarcoma, Soft Tissue; Leiomyosarcoma; Liposarcoma; Pleomorphic Liposarcoma
Keywords: sarcoma
MeSH Terms: conditions — Liposarcoma, Myxoid; Sarcoma; Leiomyosarcoma; Liposarcoma | interventions — Trabectedin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Trabectedin+Radiotherapy (Experimental): Trabectedin 1.3 or 1.5mg/m2 and radiotherapy 30Gy or 45Gy.
  Interventions: Drug: Trabectedin; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Trabectedin — Escalating or deescalating dose of 1.3 or 1.5mg/m2, i.v 24h, once every 3 weeks.
  Cohort A: unlimited cycles. Cohort B: 3 cycles. Cohort C: 3 cycles. Cohort D: cycles of trabectedin will be provided and patients will subsequently be evaluated for surgery.
  Other Names: Yondelis
Radiation: Radiotherapy — 3D conformal radiotherapy (3D-CRT) or intensity modulated radiotherapy (IMRT) providing: Cohort A: 30Gy in 10 fractions (3Gy/fraction). Cohort B: 45Gy in 25 fractions (1.8Gy/fraction). Cohort C: 45Gy in 25 fractions (1.8Gy/fraction). Cohort D: 45Gy in 25 fractions (1.8Gy/fraction).

SUMMARY:
Phase I-II trial that combines trabectedin plus radiotherapy for tumor reduction response measure in four cohorts of patients:

Cohort A: Patients with diagnosis of non-operable or unresectable or not oncologically recommended metastasectomy of limited to lung metastases soft tissue sarcoma.

Cohort B: Patients with locally advanced resectable Myxoid Liposarcoma. Cohort C: Patients with retroperitoneal and resectable soft tissue sarcoma (liposarcoma and leiomyosarcoma).

Cohort D (Phase II only): Patients with well differentiated liposarcoma and G2 dedifferentiated liposarcoma (with less than 30% dedifferentiated component).

Phase I: escalating dose of 1.3 or 1.5 mg/m2. Phase I for cohort C: de-escalating dose of 1.5 or 1.3mg/m2 Radiotherapy for cohort A: 30Gy in 10 fractions (3Gy/fraction). Radiotherapy for cohort B: 45Gy in 25 fractions (1.8Gy/fraction). Radiotherapy for cohort C: 45Gy in 25 fractions (1.8Gy/fraction).

Radiotherapy for cohort D: 45Gy in 25 fractions (1.8Gy/fraction). A translational substudy is developed to analyse different biomarkers predictive value.

Cohorts A and B are closed to recruitment in 2023.

DETAILED DESCRIPTION:
In this study investigators plan to measure tumor response (RECIST and Choi criteria) when administering trabectedin standard dose or inferior with simultaneous radiotherapy treatment. The hypothesis states that administering trabectedin at 1.3mg/m2 or ≤1.5mg/m2 plus Radiotherapy 30-45Gy shows synergic activity that turns into tumor shrinkage.

A phase I trial (dose escalation -or de-escalation for cohort C- level of 1.3 or 1.5 mg/m2) will provide the proper dose level to perform a phase II trial to measure RECIST and Choi response, progression free survival, overall survival and register safety and quality of life details.

Four cohorts are indicated for this trial:

Cohort A: Patients with diagnosis of non-operable or unresectable or not oncologically recommended metastasectomy of limited to lung metastases soft tissue sarcoma.

Cohort B: Patients with locally advanced resectable Myxoid Liposarcoma, Cohort C:Patients with retroperitoneal and resectable soft tissue sarcoma (liposarcoma and leiomyosarcoma).

Cohort D: Patients with well differentiated liposarcoma and G2 dedifferentiated liposarcoma (with less than 30% dedifferentiated component) Unlimited cycles of chemotherapy are considered to be beneficial for cohort A patients, whereas cohort B and C only 3 cycles are indicated. About radiotherapy treatment, 30Gy will be given to cohort A patients, whereas cohort B and C will receive 45Gy. TCs and MRI are selected for imaging purposes.

Phase I:

For cohorts A and B:Trabectedin at two dose escalation levels:

0 1.3 mg/m2 as a 24h I.V. infusion

1 1.5 mg/m2 as a 24h I.V. infusion

For cohort C:Trabectedin at two dose de-escalation levels:

0 1.5 mg/m2 as a 24h I.V. infusion

-1 1.3 mg/m2 as a 24h I.V. infusion

Administration of trabectedin with a portable pump, i.v infusion of 24h, in cycles of 3 weeks.

Premedication:

* 4 mg oral dexamethasone 24h and 12h before chemotherapy administration.
* 20 mg I.V. dexamethasone 30minutes before treatment.
* Ondansetron or analogue will also be given prior to trabectedin.

Pathology review, radiology review and radiotherapy review are performed to each patient.

Several biomarkers are selected to perform FFPE tumor assays in relation to prediction

ELIGIBILITY:
Cohort A: STS

Inclusion Criteria:

1. The patient must sign voluntarily the informed consent form before any study test is conducted that is not part of routine patient care.
2. Aged equal or over 18.
3. Patients must have a diagnostic of Soft Tissue Sarcoma with metastasis limited to lung, and not suitable for metastasectomy or surgery resection or not oncologically recommended metastasectomy.A centralized diagnostic will be performed, the tumor sample must be available and sent prior to inclusion.
4. Disease distribution allows meeting with normal tissue constraints of radiation therapy. Radiation oncologist must confirm this point.
5. Metastatic spread could be present in two organs at maximum (i.e. lungs and pelvic fosa).
6. Those lesions considered for radiation therapy have to be considered as target lesions as well. (i.e. in a patient with nodules in lungs, those lesions selected for radiation therapy have to include at least the target lesions)
7. It is allowed that not all the lesions will be under radiation fields. As a general rule, it will be prioritized to select, as target-irradiating lesions, those with greater increase in size and those largest lesions. It should be discouraged to irradiate pulmonary lesions with infiltration of pleural serosa.
8. Patients must have documentation of disease progression within 6 months prior to study entry.
9. The patient must have been considered eligible for systemic chemotherapy. A maximum of two previous lines for advanced/metastatic disease are allowed as long as trabectedin has not been included.
10. The following histological subtypes can be included:

    Undifferentiated pleomorphic sarcoma (previously, malignant fibrous histiocytoma) Leiomyosarcoma Angiosarcoma/ epithelial hemangioendothelioma Liposarcoma and its variants (well differentiated, dedifferentiated, myxoid/round cells, pleomorphic).

    Synovial sarcoma Fibrosarcoma and its variants (epithelial fibrosarcoma/low grade fibromyxoid sarcoma) Hemangiopericytoma/solitary fibroid tumor Neurogenic sarcoma (Malignant peripheral nerve sheath tumor, MPNST) Myxofibrosarcoma Epithelioid Sarcoma Unclassified sarcoma (spindle cell/epithelioid/pleomorphic/myxoid)
11. Measurable disease, according to RECIST V 1.1 criteria
12. Performance status ≤1 (ECOG).
13. Adequate respiratory functions: FEV1 >1L; DLco > 40% (patients with pulmonary target lesions)
14. Adequate bone marrow function (hemoglobin > 10 g/dl, leukocytes ≥ 3.000/mm3, neutrophils ≥ 1.500/mm3, platelets ≥ 100.000/mm3). Patients with plasma creatinine ≤ 1,6 mg/dl, transaminases ≤ 2.5 times the UNL, total bilirubin ≤ UNL, CPK ≤ 2.5 times UNL, alkaline phosphatase ≤ 2.5 times the UNL are acceptable. If the increase of alkaline phosphatase is > 2.5 times the UNL, then the alkaline phosphatase liver fraction and/or GGT must be ≤ UNL.
15. Men or women of child bearing potential should be using an effective method of contraception before entry into the study and throughout the same and for 6 months after ending the study. Women of childbearing potential must have a negative urine pregnancy test before study entry.
16. Normal cardiac function with a LVEF ≥ 50% by echocardiogram or MUGA.
17. It should be performed HBV and HCV serologies prior to inclusion. If HbsAg is positive it is recommended to reject the existence of replicative phase (HbaAg+, DNA VHB+). If these were positives the inclusion is not recommended, remaining at investigators' discretion the preventive treatment with lamivudine. If a potential patient is positive for anti-HCV antibodies, presence of the virus should be ruled out with a qualitative PCR, or the patient should NOT be included in the study (if a qualitative PCR cannot be performed then patient will not be able to enter the study)
18. Patient must have a Central Venous Catheter for treatment

Exclusion Criteria:

1. Previous treatment with trabectedin or previous treatment with radiotherapy (except if previous radiotherapy treatment plus planned study radiotherapy treatment allow tissues constrains)
2. Performance status ≥ 2 (ECOG).
3. Plasma bilirubin > UNL.
4. Creatinine > 1.6 mg/dL.
5. History of other neoplastic disease with less than 5 years free of disease with the exception of basal cell carcinoma or in situ cervical cancer adequately treated.
6. Severe COPD or other severe pulmonary diseases.
7. Significant cardiovascular disease (for example, dyspnea > 2 NYHA)
8. Significant systemic diseases grade 3 or higher on the NCI-CTCAE v4.03 scale, that limit patient availability, or according to investigator judgment may contribute significantly to treatment toxicity.
9. Uncontrolled bacterial, mycotic or viral infections.
10. Known positive test for infection by human immunodeficiency virus (HIV).
11. Women who are pregnant or breast-feeding.
12. Psychological, familial, social or geographic circumstances that limit the patient"s ability to comply with the protocol or informed consent.
13. Patients participating in another clinical trial or receiving any other investigational product
14. Patients who had participated in another clinical trial and/or had received any other investigational product in the last 30 days prior to inclusion.
15. Histologies other than those described in inclusion criteria.

Cohort B: ML

Inclusion criteria:

1. The patient must sign voluntarily the informed consent form before any study test is conducted that is not part of routine patient care.
2. Age ≥18 years old.
3. Pathological diagnosis of Myxoid Liposarcoma, deep located and more than 5 cm or superficial more than 10 cm. A centralized diagnostic will be performed to confirm that the patient can be included in the study.
4. Tumor must be resectable and without evidence of regional or distal spread after adequate staging procedure. Tumor must be located in limbs or superficial trunk wall.
5. Disease distribution allows meeting with normal tissue constraints of radiation therapy. Radiation oncologist must confirm this point.
6. Measurable disease, according to RECIST V 1.1 criteria
7. Performance status 0-1 (ECOG).
8. Adequate bone marrow function (hemoglobin > 10 g/dL, leukocytes ≥ 3.000/mm3, neutrophils ≥ 1.500/mm3, platelets ≥ 100.000/mm3). Patients with plasma creatinine ≤ 1,6 mg/dL, transaminases ≤ 2.5 times the UNL, total bilirubin ≤ UNL, CPK ≤ 2.5 times UNL, alkaline phosphatase ≤ 2.5 times the UNL are acceptable. If the increase of alkaline phosphatase is > 2.5 times the UNL, then the alkaline phosphatase liver fraction and/or GGT must be ≤ UNL.
9. Men or women of child bearing potential should be using an effective method of contraception before entry into the study and throughout the same and for 6 months after ending the study. Women of childbearing potential must have a negative urine pregnancy test before study entry.
10. Normal cardiac function with a LVEF ≥ 50% by echocardiogram or MUGA.
11. It should be performed HBV and HCV serologies prior to inclusion. If HbsAg is positive it is recommended to reject the existence of replicative phase (HbaAg+, DNA HBV+). If these were positives the inclusion is not recommended, remaining at investigators' discretion the preventive treatment with lamivudine. If a potential patient is positive for anti-HCV antibodies, presence of the virus should be ruled out with a qualitative PCR, or the patient should NOT be included in the study (if a qualitative PCR cannot be performed then patient will not be able to enter the study).
12. Patient may have had one previous chemotherapy line.
13. Patient must have a Central Venous Catheter for treatment.

Exclusion criteria:

1. Unresectable tumors (with limb sparing surgery)
2. More than one previous chemotherapy treatment for local disease including trabectedin.
3. Radiotherapy involving the tumoral bed.
4. Performance status ≥ 2 (ECOG).
5. Presence of metastases or lymph node involvement by the tumor.
6. Location other than limb or superficial trunk wall.
7. Plasma bilirubin > UNL.
8. Creatinine > 1.6 mg/dL.
9. History of other neoplastic disease with less than 5 years free of disease with the exception of basal cell carcinoma or in situ cervical cancer adequately treated.
10. Significant cardiovascular disease (for example, dyspnea > 2 NYHA)
11. Significant systemic diseases grade 3 or higher on the NCI-CTCAE v4.03 scale, that limit patient availability, or according to investigator judgment may contribute significantly to treatment toxicity.
12. Uncontrolled bacterial, mycotic or viral infections.
13. Known positive test for infection by human immunodeficiency virus (HIV).
14. Women who are pregnant or breast-feeding.
15. Psychological, familial, social or geographic circumstances that limit the patient"s ability to comply with the protocol or informed consent.
16. Patients who had participated in another clinical trial and/or had received any other investigational product in the last 30 days prior to inclusion.

Cohorts C and D: Retroperitoneum sarcoma

Inclusion criteria:

1. The patient must voluntarily sign the informed consent form before performing any study-specific test that is not part of the patient's usual care.
2. Aged between 18 and 75 years.
3. The following histological subtypes may be included in the cohort C:

   High grade leiomyosarcoma (G2-3), liposarcoma (G2-3), if at least 30% of the tumour is dedifferentiated, pleomorphic liposarcoma.

   The following histological subtypes may be included in the cohort D:

   Well differentiated liposarcoma (WD liposarcoma) and G2 dedifferentiated liposarcorcoma, if less than 30% of the tumour is dedifferentiated.

   A centralised diagnosis will be made to confirm that the patient can be included in the study.
4. The tumour must be located in the retroperitoneum and it must be resectable and without evidence of regional or distal spread after the appropriate staging process. This point must be confirmed by the central surgeon reviewer.
5. The location and size of the disease in the retroperitoneum must allow for compliance with radiotherapy limitations in healthy tissue. This point must be confirmed by the site's radiation oncologist and the central radiation oncologist reviewer.
6. Measurable disease according to CHOI criteria for cohort C and RECIST V 1.1 criteria for cohort D.
7. ECOG performance status 0-1.
8. Adequate haematological parameters (haemoglobin >10 g/dl, leukocytes ≥3,000/mm3, neutrophils ≥1,500/mm3, platelets ≥100,000/mm3). Patients with plasma creatinine ≤1.6 mg/dl, transaminases ≤2.5 times the ULN, total bilirubin ≤ ULN, CPK ≤2.5 times ULN, alkaline phosphatase ≤2.5 times ULN are acceptable. If the increase in alkaline phosphatase is >2.5 times the ULN, the liver fraction of alkaline phosphatase and/or GGT should be ≤ULN.
9. Fertile men or women must use an effective contraceptive method before starting the study, during the study and for 6 months following the conclusion thereof. Women of childbearing potential who participate in the study must undergo a pregnancy test before starting the study.
10. Normal cardiac function with LVEF ≥50% by echocardiogram or MUGA.
11. HBV and HCV serology must be performed before including the patient in the study. If HbsAg is positive, it is advisable to rule out a replicative phase (HbsAg*, DNA HBV+). If positive, the patient's inclusion in the trial is not recommended, and it is at the discretion of the investigator to administer preventive treatment with lamivudine. If a potential patient is positive to anti-HCV antibodies, the presence of the virus will be ruled out with a qualitative PCR, or the patient cannot be included in the study (if the qualitative PCR test cannot be performed on the patient, they cannot be included in the study).
12. Patient may have had one previous chemotherapy line (cohort D only).
13. The patient must have a central venous catheter for the administration of the treatment.

Exclusion criteria

1. Unresectable tumours.
2. Location other than the retroperitoneum.
3. Patients who have previously received systemic treatment with chemotherapy (trabectedin included). For cohort D, patients may have received one previous line of chemotherapy with any other agent.
4. Patients who underwent prior local treatment for retroperitoneal sarcoma: surgery or radiotherapy in the tumour bed.
5. ECOG performance status ≥2.
6. Presence of metastasis or lymph node involvement of the tumour.
7. Previous history of another neoplastic disease with less than 5 years free of disease except for basal cell carcinoma or properly treated in situ cervical cancer.
8. Significant cardiovascular disease (e.g. dyspnoea >2 NYHA).
9. A significant grade 3 or greater systemic disease on the NCI-CTCAE v4.03 scale, which may limit the availability of the patient or which, in the opinion of the investigator, may contribute to the toxicity caused by the study treatment.
10. Uncontrolled viral, mycotic or bacterial infections.
11. Known HIV-positive patients.
12. Pregnant or breast-feeding women.
13. Psychological, familial, social or geographical circumstances that limit the patient's ability to comply with the protocol or informed consent form.
14. Patients who have participated in another clinical trial and/or have received another investigational product in the 30 days prior to inclusion in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Estimated)
Dates: Start 2014-11 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Tumor size | every 6 weeks for 24 months
  Image tumor assessment: RECIST response for the combination of trabectedin plus radiation therapy in cohorts A and B. CHOI response for the combination of trabectedin plus radiation therapy in cohort C.
Relapse-free survival. | 5 years.
  In cohort D to improve 5-year relapse-free survival (RFS), decreasing the 5-year relapse percentage from 30% to 10% in patients with well differentiated liposarcoma with cellular component and dedifferentiated G2 retroperitoneal resected liposarcoma (20% increase in RFS).

SECONDARY OUTCOMES:
Number and grade of adverse events | every 21 days until 30 days after last dose or during 25 months
  CTCAE v4.03 adverse events registration to evaluate safety
Number of months without progression | 24 months
  Progression free survival (PFS)
Number of months alive | 24 months
  Overall survival (OS)
Tumor size | every 6 weeks during 24 months (cohort A) or every 4months during 36 months (cohort B and C)
  Image tumor assessment measured by Choi criteria.
Questionnaire | every 3 months during 24 months
  QLQ-C30 EORTC questionnaire to evaluate patient quality of life
Overall response rate (ORR) | every 6 weeks during 24 months
  Sum of complete responses, partial responses and stable diseases
relapse free survival (RFS) at 3 years (cohorts C and D) | After 3 year since last patient treatment initiation
  percentage of relapses from diagnosis at 3 years
relapse at 5 years (cohorts C and D) | After 5 years since last patient treatment initiation
  number of months without relapse from treatment initiation until 5 years.
Tumor cells response to the treatment | Week 11, at surgery
  Number of tumor necrotic cells
Predictive and prognostic biomarker | Baseline and week 11 (at surgery)
  percentage of protein and RNA expression of FAS, Ca2+ and NER pathways in tumor samples obtained at baseline and at surgery (approx week 11)

CONTACTS AND LOCATIONS:
Overall Officials: Javier Martín-Broto, MD, Principal Investigator — Jiménez Díaz Foundation University Hospital
Locations (17):
- France (2):
  - Institut Bergonié, Bordeaux
  - Centre Léon Berard, Lyon
- Italy (5):
  - Istituto Clinico Humanitas, Rozzano, Milan
  - Centro di Referimento Ocologico, Aviano
  - Istituto Ortopedico Rizzoli, Bologna
  - Candiolo Cancer Institute, Candiolo
  - Istituto Nazionale dei Tumori, Milan
- Spain (10):
  - Hospital Miguel Servet, Zaragoza, Aragon
  - Hospital Sant Pau, Barcelona, Catalonia
  - Hospital Son Espases, Palma de Mallorca, Mallorca
  - Hospital Universitario Canarias, San Cristóbal de La Laguna, Tenerife
  - Hospital Vall d'Hebrón, Barcelona
  - Hospital Puerta de Hierro, Madrid
  - Hospital Universitario Gregorio Marañón, Madrid
  - Hospital Uniersitario La Paz, Madrid
  - Jiménez Díaz Foundation University Hospital, Madrid
  - Hospital Virgen del Rocío, Seville

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vatner R, James CD, Sathiaseelan V, Bondra KM, Kalapurakal JA, Houghton PJ. Radiation therapy and molecular-targeted agents in preclinical testing for immunotherapy, brain tumors, and sarcomas: Opportunities and challenges. Pediatr Blood Cancer. 2021 May;68 Suppl 2:e28439. doi: 10.1002/pbc.28439. Epub 2020 Aug 22. PMID 32827353
- [Derived] Martin-Broto J, Hindi N, Lopez-Pousa A, Peinado-Serrano J, Alvarez R, Alvarez-Gonzalez A, Italiano A, Sargos P, Cruz-Jurado J, Isern-Verdum J, Dolado MC, Rincon-Perez I, Sanchez-Bustos P, Gutierrez A, Romagosa C, Morosi C, Grignani G, Gatti M, Luna P, Alastuey I, Redondo A, Belinchon B, Martinez-Serra J, Sunyach MP, Coindre JM, Dei Tos AP, Romero J, Gronchi A, Blay JY, Moura DS. Assessment of Safety and Efficacy of Combined Trabectedin and Low-Dose Radiotherapy for Patients With Metastatic Soft-Tissue Sarcomas: A Nonrandomized Phase 1/2 Clinical Trial. JAMA Oncol. 2020 Apr 1;6(4):535-541. doi: 10.1001/jamaoncol.2019.6584. PMID 32077895
- [Derived] Gronchi A, Hindi N, Cruz J, Blay JY, Lopez-Pousa A, Italiano A, Alvarez R, Gutierrez A, Rincon I, Sangalli C, Perez Aguiar JL, Romero J, Morosi C, Sunyach MP, Sanfilippo R, Romagosa C, Ranchere-Vince D, Dei Tos AP, Casali PG, Martin-Broto J. Trabectedin and RAdiotherapy in Soft Tissue Sarcoma (TRASTS): Results of a Phase I Study in Myxoid Liposarcoma from Spanish (GEIS), Italian (ISG), French (FSG) Sarcoma Groups. EClinicalMedicine. 2019 Mar 11;9:35-43. doi: 10.1016/j.eclinm.2019.03.007. eCollection 2019 Mar. PMID 31143880